CLINICAL TRIAL: NCT06494579
Title: A Phase 1b/2 Trial of Lamivudine in the Treatment of Relapsed/Refractory Solid Tumors Progression on Anti-PD-(L)1 Blockade
Brief Title: Lamivudine for Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Thomas Marron (Other)
Responsible Party: Sponsor-Investigator, Thomas Marron, Professor, Hematology Oncology, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-24-00614
Record Dates: First submitted 2024-06-27; First posted 2024-07-10 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Relapsed/Refractory Solid Tumors
MeSH Terms: conditions — Recurrence | interventions — Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with Relapsed Refractory Solid Tumors (Experimental): Participants with Solid Tumors which are typically treated with cancer immunotherapy (PD-1 or PD-L1 blocking antibodies) and their cancer has progressed on immunotherapy will be candidates for the trial. This is a single-arm trial.
  Interventions: Drug: Lamivudine; Drug: PD-L1 Blocker

INTERVENTIONS:
Drug: Lamivudine — Lamivudine is used in the management of human immunodeficiency virus (HIV) and Hepatitis B Virus. It is being repurposed here to assess if this can improve response to cancer immunotherapy
Drug: PD-L1 Blocker — PD-1 or PD-L1 blocking antibodies; there are around a dozen of these FDA approved for varying indications, and whatever is administered to a patient as standard of care (FDA APPROVED) will be continued in the patients and administered in combination with lamivudine.

SUMMARY:
Single arm, set dose clinical trial of Lamivudine for Relapsed Refractory Solid Tumors.

Accrual 6-24 patients, within 2 years, study completion within 3 years at Mount Sinai Health System.

Primary Objective:

For Phase 1b to determine the safety and tolerability of Lamivudine with continued PD-(L)1 blockade for patients with relapsed/refractory metastatic solid tumors that have progressed on standard PD-(L)1 blockade.

For Phase 2, to determine the effect of adding lamivudine to PD-(L)1 blocking agents in patients with relapsed/refractory solid tumors that have progressed on prior PD-(L)1 agents

Secondary Objectives (Phase 1b and 2) Assess 1) Safety and Tolerability, 2) Best overall response rate (BORR), 3) Progression-free survival (PFS), 4) Overall survival (OS) and 5) Duration of response following addition of lamivudine to standard PD-(L)1 blocking agents, 6) Disease control rate (DCR).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a pathologically confirmed diagnosis of a solid malignancy
* Patients must have progressed (clinically or radiographically) on or following prior therapy with a PD-1 or PD-L1 targeted antibody
* Patients must have exhausted or declined all standard therapies deemed to have significant clinical benefit
* Patients may have only 0 or 1 intervening lines of therapy from the prior PD-(L)1 blocking therapy
* Patient must be willing and able to provide blood samples (12 green-top tubes, roughly 100mL) at the four time points indicated in the Study Calendar.
* Age ≥ 18 years.
* ECOG 0-2. The exception will be patients carrying long term disability (such as cerebral palsy) where the disability is not acute nor progressive, and unlikely to significantly affect their response to therapy. This must be documented in screening clinic visit note by investigator.
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 3 months following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 24 consecutive months
* Ability to understand and the willingness to sign a written informed consent.
* Adequate organ and marrow function

Exclusion Criteria

* Patients who have had chemotherapy within 14 days from start of therapy.
* Patients who have had radiotherapy within 7 days from start of therapy, though exception may be made for palliative radiotherapy which is permitted at anytime, if deemed in the best interest of the patient.
* Patients may not be receiving any other investigational agents.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring antibiotics (exception is a brief (≤10days) course of antibiotics to be completed before initiation of treatment), symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Exception: Patients on chronic steroids (more than 4 weeks at stable dose) equivalent to ≤ 10mg prednisone will not be excluded.
* Has active autoimmune disease that has required systemic treatment in the past 1 year (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Exception: Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is acceptable.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.
* Known HIV positive with detectable viral load, or anyone not on stable anti-viral (HAART) regimen, or with <350 CD4+ T cells/microliter in the peripheral blood. HIV testing is not required for patients with no known history of HIV.
* Any patient already on antiretroviral therapy
* Has known Hepatitis B or active Hepatitis C (e.g., HCV RNA [qualitative] is detected). HBV and HCV testing is not required for patients with no known history of these viruses.
* History of allogeneic hematopoietic cell transplantation or solid organ transplantation.
* Receipt of a live vaccine within 30 days of planned start of study drug
* Documented allergic or hypersensitivity response to any protein therapeutics (e.g., recombinant proteins, vaccines, intravenous immune globulins, monoclonal antibodies, receptor traps). Principal investigator believes that for one or multiple reasons the patient will be unable to comply with all study visits, or if they believe the trial is not clinically in the best interest of the patient.
* History of irAE in response to prior immunotherapy that has not improved to a Grade 0 or 1; this does not include chronic conditions such as endocrinopathies which can be treated with hormone replacement therapy.
* History of interstitial lung disease (e.g., idiopathic pulmonary fibrosis, organizing pneumonia) or active, noninfectious pneumonitis attributed to prior use of cancer immunotherapy that required immune-suppressive doses of glucocorticoids to assist with management. A history of radiation pneumonitis in the radiation field is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-09-26 (Actual); Primary Completion 2026-07-28 (Estimated); Study Completion 2026-07-28 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLTs) per CTCAE Version 5.0 | Cycle 1, each cycle is 21 days
  Dose-limiting toxicity rate in the first 6 patients based on the CTCAE version 5.0. DLTs were defined as any Lamivudine-related Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE 5.0) Grade 3 or 4 adverse events.

SECONDARY OUTCOMES:
DLT of combined treatment of lamivudine and PD-(L)1 targeted therapy. | Cycle 1, each cycle is 21 days
  To determine the safety and tolerability of combined treatment of lamivudine and PD-(L)1 targeted therapy in patients with relapsed or refractory solid tumors. DLTs were defined as any treatment-related Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE 5.0) Grade 3 or 4 adverse events.
Best overall response rate (BORR). | End of study at 3 years
  Best overall response rate (BORR), defined as the percent of patients achieving a Complete Response (CR) or Partial Response (PR) on initial or subsequent imaging before initiation of subsequent line of anti-cancer therapy
Overall survival (OS) | End of study at 3 years
  Overall survival (OS): defined as the time from the first dosing of lamivudine and date of death
Progression free survival (PFS): | End of study at 3 years
  Progression free survival (PFS): defined as the time from first dosing of lamivudine to date of objectively documented progression of disease or death
Duration of response (DOR) | End of study at 3 years
  Duration of response (DOR): defined as the time between the date of first response of CR or PR to the date of first documented tumor progression or death due to any cause
Disease control rate (DCR) | End of study at 3 years
  Disease control rate (DCR): defined as percent of patients experiencing CR, PR or Stable Disease (SD) at the time of first imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Marron, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose. To achieve aims in the approved proposal. Proposals should be directed to Sponsor-Investigator at thomas.marron@mssm.edu.